CLINICAL TRIAL: NCT04308304
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Pharmacokinetics of MK-1942 Administered to Alzheimer's Disease Patients Receiving Donepezil Treatment.
Brief Title: MK-1942/Donepezil Interactions in Participants With Alzheimer's Disease (MK-1942-005)
Acronym: DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1942-005; MK-1942-005 (Other: Merck Protocol Number)
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Donepezil
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donepezil (Experimental): Participants receive Dose Level 1: 8-mg MK-1942 twice daily (BID) x 7 days (7D), Day 1 to Day 7; Dose Level 2: 15-mg MK-1942 BID x 7D, Day 8 to Day 14; Dose Level 3: 30-mg MK-1942 BID x 7D, Day 15 to Day 21; Dose Level 4: ≤50-mg MK-1942 BID x 7D (Provisional Dose Level), Day 22 to Day 28 All participants to receive Donepezil once daily.
  Interventions: Drug: MK-1942; Drug: Donepezil
- Placebo (Placebo Comparator): Placebo to MK-1942 BID x 21 [28] D All participants to receive Donepezil once daily.
  Interventions: Drug: Donepezil; Drug: Placebo

INTERVENTIONS:
Drug: MK-1942 — MK-1942 1 mg, 5 mg, and/or 10 mg capsules taken twice daily (BID) by mouth.
  Arms: Donepezil
Drug: Donepezil — Donepezil 5 mg and/or 10 mg tablets taken once daily (QD) by mouth.
Drug: Placebo — Placebo capsule matched to MK-1942 taken BID by mouth.
  Arms: Placebo

SUMMARY:
The study investigated the effects on safety and pharmacokinetics (PK) of MK-1942 and donepezil when co-administered to participants with Alzheimer's Disease with mild-to-moderate cognitive impairment stably treated with donepezil. The objectives of this study were to determine if the combination of MK-1942 with donepezil increases the incidence or severity of adverse events (AEs) previously reported for these agents alone, or results in unanticipated AEs in the patient population targeted for MK-1942 treatment. In addition, changes in the PK parameters of either MK-1942 or donepezil as a result of co-administration were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18 and ≤35 kg/m^2, inclusive.
* Is in good health based on medical history, physical examination, vital sign measures and electrocardiogram performed prior to randomization.
* Have a negative urine drug screen prior to randomization.
* Have a history of cognitive and functional decline with gradual onset and slow progression for at least one year before screening that is either corroborated or well-documented.
* Be receiving donepezil (maximum dose: ≥10-mg, ≤15-mg) for symptomatic treatment of cognitive impairment associated with Alzheimer's dementia. The dose level must be stable for at least 1 month prior to screening.
* Have a reliable and competent trial partner/caregiver who has a close relationship with the subject, has face-to-face contact at least three days a week for a minimum of six waking hours a week, and is willing to accompany the participant, if desired, to trial visits. The trial partner/caregiver should understand the nature of the trial and adhere to trial requirements (e.g., dosing, visit schedules, and nature and number of evaluations).
* Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Male participants must refrain from donating sperm PLUS agree to study guidelines regarding abstinent and/or contraception during the intervention period and for at least an additional 90 days (a spermatogenesis cycle) after the last dose of study intervention:
* A female participant is eligible to participate if she is a women of nonchildbearing potential by study criteria.

Exclusion Criteria:

* Is positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV).
* Is at imminent risk of self-harm, based on clinical interview and responses on the Columbia-Suicide Severity Rating Scale (CSSRS), or of harm to others in the opinion of the investigator.
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pretrial (screening) visit.
* Has a history of uncontrolled, clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* Candidates should not have a history of asthma, chronic obstructive pulmonary disease, urinary obstructions or gastrointestinal bleeding.
* Has a history of cancer (malignancy) exceptions for (1) Adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix or; (2) Other malignancies which have been successfully treated with appropriate follow up and therefore unlikely to recur for the duration of the study.
* Has a history of significant multiple and/or severe allergies (e.g., food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e., systemic allergic reaction) to prescription or non-prescription drugs or food.
* Has evidence of a clinically relevant or unstable psychiatric disorder, based on The Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria, including schizophrenia or other psychotic disorder, bipolar disorder, or delirium at the time of the pre-study (screening) visit, or has a history of clinically significant psychiatric disorder of the last 5 years.
* Has participated in another investigational study within 4 weeks (or 5 half-lives, whichever is greater) prior to the pre-study (screening) visit.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- United States (4):
  - Woodland Research Northwest, LLC ( Site 0004), Rogers, Arkansas
  - Velocity Clinical Research, Hallandale Beach ( Site 0002), Hallandale, Florida
  - iResearch Atlanta ( Site 0005), Decatur, Georgia
  - ICON ( Site 0003), Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female adult (≥50 to ≤85 years of age) participants with Alzheimer's disease (AD) and mild-to-moderate cognitive impairment were enrolled at 4 study centers in the United States.
Groups:
- MK-1942 AD: Participants with AD receive donepezil 10 mg to 15 mg once daily (QD), and MK-1942 twice daily (BID), for 28 days. Doses of MK-1942 were 8 mg (Week 1), 15 mg (Week 2), 30 mg (Week 3) and 50 mg (Week 4).
- Placebo + Donepezil AD: Participants with AD receive donepezil 10 mg to 15 mg QD, and placebo BID, for 28 days.
Period: Overall Study
Arm/Group | MK-1942 AD | Placebo + Donepezil AD
Started | 22 | 5
Completed | 17 | 5
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-1942 AD | Placebo + Donepezil AD | Total
Number analyzed (Participants) | 22 | 5 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (5.5) | 69.4 (2.6) | 69.2 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 12
  Male | 12 | 3 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 4 | 23
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 0 | 7
  White | 15 | 5 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ≥1 Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to Day 42
Population: All participants who received ≥1 dose of study treatment are included.
Measure: Count of Participants; unit: Participants
Groups:
- MK-1942 8 mg + Donepezil AD: Participants with AD received MK-1942 8 mg + donepezil during Week 1.
- MK-1942 15 mg + Donepezil AD: Participants with AD received MK-1942 15 mg + donepezil during Week 2.
- MK-1942 30 mg + Donepezil AD: Participants with AD received MK-1942 30 mg + donepezil during Week 3.
- MK-1942 50 mg + Donepezil AD: Participants with AD received MK-1942 50 mg + donepezil during Week 4.
Arm/Group | MK-1942 8 mg + Donepezil AD | MK-1942 15 mg + Donepezil AD | MK-1942 30 mg + Donepezil AD | MK-1942 50 mg + Donepezil AD | Placebo + Donepezil AD
Number analyzed (Participants) | 22 | 19 | 15 | 15 | 5
Participants | 13 | 4 | 4 | 5 | 4

2. Primary Outcome: Number of Participants Discontinuing From Study Therapy Due to an Adverse Event (AE)
Description: as for outcome 1
Time Frame: Up to Day 28
Population: All participants who received ≥1 dose of study treatment are included.
Measure: Count of Participants; unit: Participants
Groups:
- MK-1942 8 mg AD: Participants with AD received MK-1942 8 mg + donepezil during Week 1.
- MK-1942 15 mg AD: Participants with AD received MK-1942 15 mg + donepezil during Week 2.
- MK-1942 30 mg AD: Participants with AD received MK-1942 30 mg + donepezil during Week 3.
- MK-1942 50 mg AD: Participants with AD received MK-1942 50 mg + donepezil during Week 4.
- Placebo AD: Participants with AD receive donepezil 10 mg to 15 mg QD, and placebo BID, for 28 days.
Arm/Group | MK-1942 8 mg AD | MK-1942 15 mg AD | MK-1942 30 mg AD | MK-1942 50 mg AD | Placebo AD
Number analyzed (Participants) | 22 | 19 | 15 | 15 | 5
Participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in 12-Lead Electrocardiogram (ECG) Findings
Description: The number of participants with clinically significant 12-lead ECGs is presented. Recordings were made throughout the study, with the participant in a semi-recumbent position having rested in this position for at least 10 minutes beforehand.
Time Frame: Up to Day 28
Population: All participants who received ≥1 dose of study treatment are included.
Measure: Count of Participants; unit: Participants
Groups:
- MK-1942 8 mg: Participants received MK-1942 8 mg + donepezil during Week 1.
- MK-1942 15 mg: Participants received MK-1942 15 mg + donepezil during Week 2.
- MK-1942 30 mg: Participants received MK-1942 30 mg + donepezil during Week 3.
- MK-1942 50 mg: Participants received MK-1942 50 mg + donepezil during Week 4.
Arm/Group | MK-1942 8 mg | MK-1942 15 mg | MK-1942 30 mg | MK-1942 50 mg | Placebo AD
Number analyzed (Participants) | 22 | 19 | 15 | 15 | 5
Participants | 1 | 0 | 0 | 0 | 1

4. Primary Outcome: Number of Participants With Abnormal (Impaired) Results on Targeted Neurological Exams
Description: The number of participants with abnormal (impaired) results on targeted neurological exams will be presented. The targeted neurological exam contains Modules 1, 2 and 5 of the general examination, focusing on arousal, cranial nerve function, and gait and will be administered several times throughout the treatment period starting on Day 1 up until Day 29. The number of participants with abnormal (impaired) results on targeted neurological exams will be reported. Each exam will be graded as Normal or Impaired with the abnormality described.
Time Frame: Up to 29 days
Population: All participants who received ≥1 dose of study treatment are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1942 8 mg | MK-1942 15 mg | MK-1942 30 mg | MK-1942 50 mg | Placebo AD
Number analyzed (Participants) | 22 | 19 | 15 | 15 | 5
Participants | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Who Reported Suicidal Ideation and/or Behavior on Study Based on Responses to the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The number of participants with suicidality using the C-SSRS is presented. The C-SSR will be used in this study only for the purpose of safety monitoring by measuring the incidence of different types of suicidality categories during treatment. C-SSRS assessment will be based upon a clinician's interpretation of the participant's responses to the C-SSRS questions, not by a numbered scale. Suicidal ideation and/or behaviors identified on the C-SSRS may not be considered an adverse event, based on the investigator's judgment. Participants who report at least one occurrence of suicidal behavior or suicidal ideation will be counted as having experienced suicidality. Suicidal behavior includes suicide attempt, aborted attempt, interrupted attempt, or preparatory behavior. Suicidal ideation include a wish to die or active suicidal thought with or without method, intent or plan.
Time Frame: Up to 42 days
Population: All participants who received ≥1 dose of study treatment are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1942 8 mg | MK-1942 15 mg | MK-1942 30 mg | MK-1942 50 mg | Placebo AD
Number analyzed (Participants) | 22 | 19 | 15 | 15 | 5
Participants | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Change From Baseline in Heart Rate (HR)
Description: The mean change from baseline in HR is presented. Change in HR was determined the first day of treatment with a new dose of MK-1942. A negative value indicates a decrease in HR relative to baseline, and a positive value indicates an increase.
Time Frame: Baseline (Day -1) and Days 1, 8, 15, and 22: 2 hours postdose
Population: All participants who received ≥1 dose of study treatment are included.
Measure: Mean (Standard Error); unit: beats/min
Arm/Group | MK-1942 8 mg | MK-1942 15 mg | MK-1942 30 mg | MK-1942 50 mg | Placebo AD
Number analyzed (Participants) | 22 | 19 | 15 | 15 | 5
beats/min | -2.27 (1.25) | 2.56 (1.65) | 6.14 (2.27) | 0.21 (2.81) | -4.53 (1.06)

7. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP)
Description: The mean change from baseline in SBP is presented. Change in SBP was determined the first day of treatment with a new dose of MK-1942. Negative values represent a decrease in SBP relative to baseline, and positive values represent an increase.
Time Frame: Baseline (Day -1) and Days 1, 8, 15, and 22: 2 hours postdose
Population: All participants who received ≥1 dose of study treatment are included.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | MK-1942 8 mg | MK-1942 15 mg | MK-1942 30 mg | MK-1942 50 mg | Placebo AD
Number analyzed (Participants) | 22 | 19 | 15 | 15 | 5
mmHg | 2.48 (2.08) | -0.15 (2.59) | 0.88 (2.09) | 1.45 (2.19) | 5.93 (4.00)

8. Primary Outcome: Mean Change From Baseline in Diastolic Blood Pressure (DBP)
Description: The mean change from baseline in DBP is presented. Change in DBP was determined the first day of treatment with a new dose of MK-1942. Negative values represent a decrease in DBP relative to baseline, and positive values represent an increase.
Time Frame: Baseline (Day -1) and Days 1, 8, 15, and 22: 2 hours postdose
Population: All participants who received ≥1 dose of study treatment are included.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | MK-1942 8 mg | MK-1942 15 mg | MK-1942 30 mg | MK-1942 50 mg | Placebo AD
Number analyzed (Participants) | 22 | 19 | 15 | 15 | 5
mmHg | -0.95 (0.93) | 0.56 (2.01) | 1.17 (1.51) | 0.10 (1.39) | -1.73 (3.36)

9. Primary Outcome: Number of Participants With Abnormal Clinical Chemistry Test Results Reported as Adverse Events
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants with abnormal chemistry-related AEs is reported.
Time Frame: Up to 42 days
Population: All participants who received ≥1 dose of study treatment are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1942 8 mg | MK-1942 15 mg | MK-1942 30 mg | MK-1942 50 mg | Placebo AD
Number analyzed (Participants) | 22 | 19 | 15 | 15 | 5
Participants | 1 | 0 | 0 | 1 | 0

10. Primary Outcome: Number of Participants With Abnormal Clinical Hematology Test Results Reported as Adverse Events
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants with abnormal hematology-related AEs is reported.
Time Frame: Up to 42 days
Population: All participants who received ≥1 dose of study treatment are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1942 8 mg | MK-1942 15 mg | MK-1942 30 mg | MK-1942 50 mg | Placebo AD
Number analyzed (Participants) | 22 | 19 | 15 | 15 | 5
Participants | 0 | 1 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Abnormal Urinalysis Results Reported as Adverse Events
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants with an abnormal urinalysis results AE is reported.
Time Frame: Up to 42 days
Population: All participants who received ≥1 dose of study treatment are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1942 8 mg | MK-1942 15 mg | MK-1942 30 mg | MK-1942 50 mg | Placebo AD
Number analyzed (Participants) | 22 | 19 | 15 | 15 | 5
Participants | 10 | 0 | 0 | 0 | 0

12. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Dosing to 12 Hours Postdose (AUC0-12) of MK-1942
Description: AUC0-12 is reported for the first day of treatment of each MK-1942 dose.
Time Frame: Days 1, 7, 14, and 21 (morning dose only): predose and 0.5, 1, 2, 3, 4, 6, and 12 hours postdose
Population: A subset of treated participants who complied with the protocol sufficiently to ensure the data are likely to reflect the underlying scientific model, are included. In addition, healthy control participant data is from study MK-1942-004.
Measure: Least Squares Mean (95% Confidence Interval); unit: hr*nmol/L
Groups:
- MK-1942 30 mg + Donepezil AD: Participants received MK-1942 30 mg + donepezil during Week 3.
- MK-1942 50 mg + Donepezil AD: Participants received MK-1942 50 mg + donepezil during Week 4.
Arm/Group | MK-1942 8 mg + Donepezil AD | MK-1942 15 mg + Donepezil AD | MK-1942 30 mg + Donepezil AD | MK-1942 50 mg + Donepezil AD
Number analyzed (Participants) | 18 | 17 | 15 | 15
hr*nmol/L | 1760 [1390 to 2240] | 3580 [2860 to 4490] | 6650 [5330 to 8280] | 11600 [9110 to 14700]
Statistical Analysis 1: Comparison: MK-1942 8 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 Alone PK; Geometric Mean Ratio (GMR) = 0.69, 90% CI 2-sided [0.55 to 0.86]
Statistical Analysis 2: Comparison: MK-1942 15 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 Alone PK; GMR = 0.66, 95% CI 2-sided [0.53 to 0.82]
Statistical Analysis 3: Comparison: MK-1942 30 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 Alone PK; GMR = 0.74, 95% CI 2-sided [0.55 to 1.00]
Statistical Analysis 4: Comparison: MK-1942 50 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 PK Alone; GMR = 0.77, 95% CI 2-sided [0.56 to 1.05]

13. Secondary Outcome: AUC From Dosing to 24 Hours Postdose (AUC0-24) of MK-1942
Description: AUC0-24 is reported for the first day of treatment of each MK-1942 dose. Due to twice daily dosing, AUC0-24 was calculated as "AUC0-24 = AUC0-12 x 2".
Time Frame: Days 1, 7, 14, and 21 (morning dose only): predose and 0.5, 1, 2, 3, 4, 6, and 12 hours postdose
Population: as for outcome 12
Measure: Least Squares Mean (95% Confidence Interval); unit: hr*nmol/L
Arm/Group | MK-1942 8 mg + Donepezil AD | MK-1942 15 mg + Donepezil AD | MK-1942 30 mg + Donepezil AD | MK-1942 50 mg + Donepezil AD
Number analyzed (Participants) | 18 | 17 | 15 | 15
hr*nmol/L | 3530 [2790 to 4470] | 7160 [5710 to 8970] | 13330 [10700 to 16600] | 23200 [18200 to 29500]
Statistical Analysis 1: Comparison: MK-1942 8 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 Alone PK; Geometric Mean Ratio (GMR) = 0.69, 90% CI 2-sided [0.55 to 0.86]
Statistical Analysis 2: Comparison: MK-1942 15 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 Alone PK; GMR = 0.66, 95% CI 2-sided [0.53 to 0.82]
Statistical Analysis 3: Comparison: MK-1942 30 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 Alone PK; GMR = 0.74, 95% CI 2-sided [0.55 to 1.00]
Statistical Analysis 4: Comparison: MK-1942 50 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 PK Alone; GMR = 0.77, 95% CI 2-sided [0.56 to 1.05]

14. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MK-1942
Description: Cmax is reported for the first day of treatment of each MK-1942 dose.
Time Frame: Days 1, 7, 14, and 21 (morning dose only): predose and 0.5, 1, 2, 3, 4, 6, and 12 hours postdose
Population: as for outcome 12
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | MK-1942 8 mg + Donepezil AD | MK-1942 15 mg + Donepezil AD | MK-1942 30 mg + Donepezil AD | MK-1942 50 mg + Donepezil AD
Number analyzed (Participants) | 18 | 17 | 15 | 15
nmol/L | 239 [184 to 310] | 477 [371 to 613] | 876 [731 to 1050] | 1360 [1080 to 1720]
Statistical Analysis 1: Comparison: MK-1942 8 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 Alone PK; Geometric Mean Ratio (GMR) = 0.67, 90% CI 2-sided [0.52 to 0.87]
Statistical Analysis 2: Comparison: MK-1942 15 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 Alone PK; GMR = 0.68, 95% CI 2-sided [0.52 to 0.87]
Statistical Analysis 3: Comparison: MK-1942 30 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 Alone PK; GMR = 0.79, 95% CI 2-sided [0.59 to 1.06]
Statistical Analysis 4: Comparison: MK-1942 50 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 PK Alone; GMR = 0.74, 95% CI 2-sided [0.51 to 1.08]

15. Secondary Outcome: Trough Plasma Concentration (Ctrough) of MK-1942
Description: Ctrough is reported for the first day of treatment of each MK-1942 dose. Data from healthy elderly participants used for statistical analyses are unpublished findings from study MK-1942-004.
Time Frame: Days 1, 7, 14, and 21 (morning dose only): predose and 0.5, 1, 2, 3, 4, 6, and 12 hours postdose
Population: as for outcome 12
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | MK-1942 8 mg + Donepezil AD | MK-1942 15 mg + Donepezil AD | MK-1942 30 mg + Donepezil AD | MK-1942 50 mg + Donepezil AD
Number analyzed (Participants) | 18 | 17 | 15 | 15
nmol/L | 101 [79.7 to 127] | 228 [188 to 277] | 386 [282 to 527] | 693 [528 to 910]
Statistical Analysis 1: Comparison: MK-1942 8 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 Alone PK; Geometric Mean Ratio (GMR) = 0.62, 90% CI 2-sided [0.48 to 0.80]
Statistical Analysis 2: Comparison: MK-1942 15 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 Alone PK; GMR = 0.67, 95% CI 2-sided [0.55 to 0.81]
Statistical Analysis 3: Comparison: MK-1942 30 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 Alone PK; GMR = 0.68, 95% CI 2-sided [0.49 to 0.93]
Statistical Analysis 4: Comparison: MK-1942 50 mg + Donepezil AD; 'MK-1942 Alone PK' are unpublished data from MK-1942-004; Test type: Other — MK-1942 + Donepezil PK / MK-1942 PK Alone; GMR = 0.72, 95% CI 2-sided [0.54 to 0.98]

16. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of MK-1942
Description: Tmax is reported for the first day of treatment of each MK-1942 dose.
Time Frame: Days 1, 7, 14, and 21 (morning dose only): predose and 0.5, 1, 2, 3, 4, 6, and 12 hours postdose
Population: as for outcome 12
Measure: Median (Full Range); unit: Hours
Arm/Group | MK-1942 8 mg + Donepezil AD | MK-1942 15 mg + Donepezil AD | MK-1942 30 mg + Donepezil AD | MK-1942 50 mg + Donepezil AD
Number analyzed (Participants) | 18 | 17 | 15 | 15
Hours | 1.97 [0.93 to 3.00] | 1.98 [0.43 to 3.00] | 2.00 [1.00 to 5.95] | 2.00 [1.93 to 3.08]

17. Secondary Outcome: Apparent Terminal Plasma Half-Life (t½) of MK-1942
Description: t½ is reported for MK-1942 50 mg.
Time Frame: Day 21 (morning dose only): predose and 0.5, 1, 2, 3, 4, 6, and 12 hours postdose
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | MK-1942 50 mg + Donepezil AD
Number analyzed (Participants) | 15
Hours | 26.7 (27.7)

18. Secondary Outcome: Apparent Clearance at Steady-state (CLss/F) of MK-1942
Description: CLss/F is reported for MK-1942 50 mg.
Time Frame: Day 21 (morning dose only): predose and 0.5, 1, 2, 3, 4, 6, and 12 hours postdose
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | MK-1942 50 mg + Donepezil AD
Number analyzed (Participants) | 15
L/h | 11.7 (45.5)

19. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vzss/F) of MK-1942
Description: Vzss/F is reported for MK-1942 50 mg.
Time Frame: Day 21 (morning dose only): predose and 0.5, 1, 2, 3, 4, 6, and 12 hours postdose
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | MK-1942 50 mg + Donepezil AD
Number analyzed (Participants) | 15
Liters | 449 (41.1)

20. Secondary Outcome: AUC0-24 of Donepezil
Description: AUC0-24 is reported for donepezil 10 mg alone (Day -1) or with MK-1942 50 mg (Day 28). Due to twice daily dosing, AUC0-24 was calculated as "AUC0-12 x 2".
Time Frame: Days 1, 7, 14, and 21 (morning dose only): predose and 0.5, 1, 2, 3, 4, 6, and 12 hours postdose
Population: A subset of treated participants who complied with the protocol sufficiently to ensure the data are likely to reflect the underlying scientific model, are included. The same participant's data are used for Day -1 and Day 28 when available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Donepezil Day -1: Participants received donepezil 10 mg alone (Day -1) or with MK-1942 50 mg (Day 28).
- Donepezil Day 28: Participants received donepezil in combination with MK-1942 for 28 days.
Arm/Group | Donepezil Day -1 | Donepezil Day 28
Number analyzed (Participants) | 20 | 15
hr*ng/mL | 606 (66.4) | 919 (44.4)
Statistical Analysis 1: Comparison: Donepezil Day -1 vs Donepezil Day 28; Test type: Other — Donepezil Accumulation Ratio (Day 28/Day -1); Geometric mean = 1.34, Standard Error of Mean 52.4

21. Secondary Outcome: Cmax of Donepezil
Description: Cmax is reported for donepezil 10 mg alone (Day -1) or with MK-1942 50 mg (Day 28).
Time Frame: Days 1, 7, 14, and 21 (morning dose only): predose and 0.5, 1, 2, 3, 4, 6, and 12 hours postdose
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Donepezil Day -1 | Donepezil Day 28
Number analyzed (Participants) | 20 | 15
ng/mL | 37.9 (56.4) | 53.3 (42.2)
Statistical Analysis 1: Comparison: Donepezil Day -1 vs Donepezil Day 28; Test type: Other — Donepezil Accumulation Ratio (Day 28/Day -1); Geometric mean = 1.22, Standard Error of Mean 52.4

22. Secondary Outcome: Ctrough of Donepezil
Description: Ctrough is reported for donepezil 10 mg alone (Day -1) or with MK-1942 50 mg (Day 28).
Time Frame: Days 1, 7, 14, and 21 (morning dose only): predose and 0.5, 1, 2, 3, 4, 6, and 12 hours postdose
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Donepezil Day -1 | Donepezil Day 28
Number analyzed (Participants) | 20 | 15
ng/mL | 20.1 (72.7) | 31.8 (52.5)
Statistical Analysis 1: Comparison: Donepezil Day -1 vs Donepezil Day 28; Test type: Other — Donepezil Accumulation Ratio (Day 28/Day -1); Geometric mean = 1.46, Standard Error of Mean 60.8

23. Secondary Outcome: Tmax of Donepezil
Description: Tmax is reported for donepezil 10 mg alone (Day -1) or with MK-1942 50 mg (Day 28).
Time Frame: Days 1, 7, 14, and 21 (morning dose only): predose and 0.5, 1, 2, 3, 4, 6, and 12 hours postdose
Population: as for outcome 20
Measure: Median (Full Range); unit: Hours
Arm/Group | Donepezil Day -1 | Donepezil Day 28
Number analyzed (Participants) | 20 | 15
Hours | 2.05 [0.00 to 4.00] | 2.03 [1.00 to 3.95]

ADVERSE EVENTS:
Time Frame: Up to 42 days
Description: All participants who received ≥1 dose of study treatment are included. Safety is reported according to MK-1942 dose or placebo treatment received.
Groups:
- MK-1942 8 mg BID 7 Days: Participants received MK-1942 8 mg + donepezil during Week 1.
- MK-1942 15 mg BID 7 Days: Participants received MK-1942 15 mg + donepezil during Week 2.
- MK-1942 30 mg Bid 7D: Participants received MK-1942 30 mg + donepezil during Week 3.
- MK-1942 50 mg BID & Days: Participants received MK-1942 50 mg + donepezil during Week 4.
- MK-1942 Total: Participants received MK-1924 8 mg, 15 mg, 30 mg, and 50 mg during Weeks 1, 2, 3, and 4, respectively.
- Placebo Bid: Participants received placebo + donepezil for 7 days.
Arm/Group | MK-1942 8 mg BID 7 Days | MK-1942 15 mg BID 7 Days | MK-1942 30 mg Bid 7D | MK-1942 50 mg BID & Days | MK-1942 Total | Placebo Bid
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/19 | 0/15 | 0/15 | 0/22 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/19 | 0/15 | 0/15 | 0/22 | 0/5
Other Adverse Events (participants affected / at risk) | 13/22 | 4/19 | 4/15 | 5/15 | 18/22 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1942 8 mg BID 7 Days (N=22) | MK-1942 15 mg BID 7 Days (N=19) | MK-1942 30 mg Bid 7D (N=15) | MK-1942 50 mg BID & Days (N=15) | MK-1942 Total (N=22) | Placebo Bid (N=5)
Scleral hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scleritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0) | 2 (3) | 7 (9) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site injury (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram T wave biphasic (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 3 (4) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT04308304/Prot_SAP_000.pdf